CLINICAL TRIAL: NCT03805659
Title: High-Definition Transcranial Direct Current Stimulation (HD-tDCS) in Logopenic Variant Primary Progressive Aphasia (lvPPA): Effects on Language and Neural Mechanisms
Brief Title: HDtDCS in Logopenic Variant PPA: Effects on Language and Neural Mechanisms
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medical College of Wisconsin (Other)
Responsible Party: Principal Investigator, Elias Granadillo Deluque, Assistant Professor, Medical College of Wisconsin
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: PRO00032037
Record Dates: First submitted 2018-12-27; First posted 2019-01-16 (Actual); Results first posted 2024-06-11 (Actual); Last update posted 2024-06-11 (Actual); Status verified 2024-05

CONDITIONS: Primary Progressive Aphasia
Keywords: Adult; Primary Progressive Aphasia; High-definition Transcranial Direct Current Stimulation; HD-tDCS; Language; Logopenic; Magnetic Resonance Imaging; MRI; Magnetoencephalography; MEG; Brain; Aphasia
MeSH Terms: conditions — Aphasia, Primary Progressive; Language; Aphasia

STUDY DESIGN:
Intervention Model Description: This is a randomized, double-blind, sham-controlled trial in which stimulation or sham will be administered to 20 subjects over the age of 45 years, with the order of treatments counterbalanced in a within-subject crossover design. Stimulation and sham sessions last 20 minutes and occur for 10 days over a 2-week period.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: An unblinded member of the study team will randomize participants to the treatment conditions. Study Group assignment will be based on random number generation (in blocks of 4) followed by the creation of numbered envelopes.
  Participants and the study team members involved in language training, tDCS delivery, and assessment of outcomes will be blind to the treatment received.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- HD-tDCS, then Sham (Experimental): Subjects receive High Dose transcranial Direct Current Stimulation (HD-tDCS) lasting 20 minutes at an electric current intensity of up to 2mA in the left posterior temporo-parietal cortex (TPC). Stimulation sessions are delivered once a day (QD) for a total of 10 sessions over 2 weeks (Monday-Friday). After a washout period of 16 weeks, subjects receive Sham sessions (no electric current) once a day (QD) for a total of 10 sessions over 2 weeks (Monday-Friday).
  Interventions: Device: HD-tDCS; Device: Sham
- Sham, then HD-tDCS (Experimental): Subjects receive Sham sessions (no electric current) once a day (QD) for a total of 10 sessions over 2 weeks (Monday-Friday). After a washout period of 16 weeks, subjects receive High Dose transcranial Direct Current Stimulation (HD-tDCS) lasting 20 minutes at an electric current intensity of up to 2mA in the left posterior temporo-parietal cortex (TPC). Stimulation sessions are delivered once a day (QD) for a total of 10 sessions over 2 weeks (Monday-Friday).
  Interventions: Device: HD-tDCS; Device: Sham

INTERVENTIONS:
Device: HD-tDCS — High-Dose transcranial Direct Current Stimulation
  Other Names: Soterix MXN-9 High-Definition stimulator
Device: Sham — Sham sessions (no electric current)

SUMMARY:
This study aims to evaluate the effectiveness of a therapy called High-Definition Transcranial Direct Current Stimulation (HD-tDCS) for the treatment of the language deficits experienced by people with a type of Primary Progressive Aphasia. This study uses a combination of brain imaging, language assessment, language training sessions, and HD-tDCS therapy as well as placebo therapy sessions.

DETAILED DESCRIPTION:
The logopenic variant of Primary Progressive Aphasia (lvPPA) is an untreatable neurodegenerative disorder that is often referred to as the 'language form' of Alzheimer's Disease (AD). Transcranial Direct Current Stimulation (tDCS) has emerged as a safe and potentially effective tool that appears to enhance language production when delivered during language training. This technology provides a critical opportunity to conduct disease intervention.

In this study, the investigators will test the hypothesis that High-Definition tDCS (HD-tDCS) will improve performance on language tasks by increasing functional connectivity and by regulating abnormal neuronal oscillatory patterns. The rationale for this project is that a determination of the therapeutic efficacy and the associated neural mechanisms of HD-tDCS in lvPPA is likely to offer a scientific framework whereby new stimulation parameters, conditions, and target sites can be deciphered.

This study will test the hypothesis that HD-tDCS will improve performance on language tasks by increasing functional connectivity and by regulating abnormal neuronal oscillatory patterns. The language performance and functional connectivity changes will be determined in a randomized, double-blind, sham-controlled crossover manner, in which a stimulation of up to 2mA in the targeted cortical tissue or sham is administered to 20 lvPPA subjects age 45 years and older. The order of treatments is counterbalanced in a within-subject crossover design. In brief, study participants will receive sham during one treatment period and stimulation during the other treatment period.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with language variant Primary Progressive Aphasia (lvPPA) subtype, defined as either clinical lvPPA or imaging-supported lvPPA in accordance with the most recent diagnostic criteria (Mesulam., 2001; Gorno-Tempini et al., 2011).
* Fluent in English.
* 45 years of age or older.
* Structural brain MRI performed within 3 years prior to enrollment.

Exclusion Criteria:

* Severe cognitive, auditory or visual impairments that would preclude cognitive testing.
* Presence of major untreated or unstable psychiatric disease.
* A chronic medical condition that is not treated or is unstable.
* The presence of cardiac stimulators or pacemakers.
* Any metal implants in the skull
* Contraindications to MRI
* History of seizures
* History of dyslexia or other developmental learning disabilities.

Min Age: 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2020-02-24 (Actual); Primary Completion 2022-05-18 (Actual); Study Completion 2022-05-18 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Elias Granadillo, Principal Investigator — The Medical College of Wisconsin
Locations (1):
- The Medical College of Wisconsin, Milwaukee, Wisconsin, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Tippett DC, Hillis AE, Tsapkini K. Treatment of Primary Progressive Aphasia. Curr Treat Options Neurol. 2015 Aug;17(8):362. doi: 10.1007/s11940-015-0362-5. PMID 26062526
- [Background] Rogalski E, Cobia D, Harrison TM, Wieneke C, Weintraub S, Mesulam MM. Progression of language decline and cortical atrophy in subtypes of primary progressive aphasia. Neurology. 2011 May 24;76(21):1804-10. doi: 10.1212/WNL.0b013e31821ccd3c. PMID 21606451
- [Background] Abel S, Weiller C, Huber W, Willmes K, Specht K. Therapy-induced brain reorganization patterns in aphasia. Brain. 2015 Apr;138(Pt 4):1097-112. doi: 10.1093/brain/awv022. Epub 2015 Feb 15. PMID 25688082
- [Background] Villamar MF, Volz MS, Bikson M, Datta A, Dasilva AF, Fregni F. Technique and considerations in the use of 4x1 ring high-definition transcranial direct current stimulation (HD-tDCS). J Vis Exp. 2013 Jul 14;(77):e50309. doi: 10.3791/50309. PMID 23893039
- [Background] Meyer AM, Snider SF, Campbell RE, Friedman RB. Phonological short-term memory in logopenic variant primary progressive aphasia and mild Alzheimer's disease. Cortex. 2015 Oct;71:183-9. doi: 10.1016/j.cortex.2015.07.003. Epub 2015 Jul 16. PMID 26232551
- [Background] Pillay SB, Stengel BC, Humphries C, Book DS, Binder JR. Cerebral localization of impaired phonological retrieval during rhyme judgment. Ann Neurol. 2014 Nov;76(5):738-46. doi: 10.1002/ana.24266. Epub 2014 Sep 19. PMID 25164766
- [Background] Gorno-Tempini ML, Brambati SM, Ginex V, Ogar J, Dronkers NF, Marcone A, Perani D, Garibotto V, Cappa SF, Miller BL. The logopenic/phonological variant of primary progressive aphasia. Neurology. 2008 Oct 14;71(16):1227-34. doi: 10.1212/01.wnl.0000320506.79811.da. Epub 2008 Jul 16. PMID 18633132
- [Background] Dancause N, Barbay S, Frost SB, Plautz EJ, Chen D, Zoubina EV, Stowe AM, Nudo RJ. Extensive cortical rewiring after brain injury. J Neurosci. 2005 Nov 2;25(44):10167-79. doi: 10.1523/JNEUROSCI.3256-05.2005. PMID 16267224
- [Background] Sonty SP, Mesulam MM, Weintraub S, Johnson NA, Parrish TB, Gitelman DR. Altered effective connectivity within the language network in primary progressive aphasia. J Neurosci. 2007 Feb 7;27(6):1334-45. doi: 10.1523/JNEUROSCI.4127-06.2007. PMID 17287508
- [Background] Datta A, Bansal V, Diaz J, Patel J, Reato D, Bikson M. Gyri-precise head model of transcranial direct current stimulation: improved spatial focality using a ring electrode versus conventional rectangular pad. Brain Stimul. 2009 Oct;2(4):201-7, 207.e1. doi: 10.1016/j.brs.2009.03.005. PMID 20648973
- [Background] Datta A, Truong D, Minhas P, Parra LC, Bikson M. Inter-Individual Variation during Transcranial Direct Current Stimulation and Normalization of Dose Using MRI-Derived Computational Models. Front Psychiatry. 2012 Oct 22;3:91. doi: 10.3389/fpsyt.2012.00091. eCollection 2012. PMID 23097644
- [Background] Muthalib M, Besson P, Rothwell J, Perrey S. Focal Hemodynamic Responses in the Stimulated Hemisphere During High-Definition Transcranial Direct Current Stimulation. Neuromodulation. 2018 Jun;21(4):348-354. doi: 10.1111/ner.12632. Epub 2017 Jul 17. PMID 28714545
- [Background] Edwards D, Cortes M, Datta A, Minhas P, Wassermann EM, Bikson M. Physiological and modeling evidence for focal transcranial electrical brain stimulation in humans: a basis for high-definition tDCS. Neuroimage. 2013 Jul 1;74:266-75. doi: 10.1016/j.neuroimage.2013.01.042. Epub 2013 Jan 28. PMID 23370061
- [Background] Richardson J, Datta A, Dmochowski J, Parra LC, Fridriksson J. Feasibility of using high-definition transcranial direct current stimulation (HD-tDCS) to enhance treatment outcomes in persons with aphasia. NeuroRehabilitation. 2015;36(1):115-26. doi: 10.3233/NRE-141199. PMID 25547776
- [Background] Kuo HI, Bikson M, Datta A, Minhas P, Paulus W, Kuo MF, Nitsche MA. Comparing cortical plasticity induced by conventional and high-definition 4 x 1 ring tDCS: a neurophysiological study. Brain Stimul. 2013 Jul;6(4):644-8. doi: 10.1016/j.brs.2012.09.010. Epub 2012 Oct 13. PMID 23149292
- [Background] Hogeveen J, Grafman J, Aboseria M, David A, Bikson M, Hauner KK. Effects of High-Definition and Conventional tDCS on Response Inhibition. Brain Stimul. 2016 Sep-Oct;9(5):720-729. doi: 10.1016/j.brs.2016.04.015. Epub 2016 Apr 22. PMID 27198577
- [Derived] Granadillo ED, Fellmeth M, Youssofzadeh V, Heffernan J, Shah-Basak PP, Pillay SB, Ustine C, Kraegel P, Schold S, Mueller KD, Ikonomidou C, Okonkwo O, Raghavan M, Binder JR. Behavioral and neural effects of temporoparietal high-definition transcranial direct current stimulation in logopenic variant primary progressive aphasia: a preliminary study. Front Psychol. 2025 Feb 25;16:1492447. doi: 10.3389/fpsyg.2025.1492447. eCollection 2025. PMID 40070907

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 6 patients were screened for eligibility between 02/24/2020 and 05/18/2022.
Pre-assignment Details: 5 of 6 subjects were randomized. 1 subject withdrew themselves prior to starting baseline procedures.
Period: Overall Study
Arm/Group | HD-tDCS, Then Sham | Sham, Then HD-tDCS
Started | 2 | 3
First Intervention (2 Weeks) | 2 | 2 (1 subject withdrew due to ongoing medical conditions unrelated to study participation)
Assessment 1 Cognitive Testing (8 Weeks After First Intervention) | 2 | 2
Washout (16 Weeks) | 2 | 2
Second Intervention (2 Weeks) | 2 | 2
Assessment 2 Cognitive Testing (8 Weeks After Intervention) | 2 | 2
Completed | 2 | 2
Not Completed | 0 | 1
Not completed — Withdrawal by Subject | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | HD-tDCS, Then Sham | Sham, Then HD-tDCS | Total
Number analyzed (Participants) | 2 | 3 | 5
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 1 | 1 | 2
  >=65 years | 1 | 2 | 3
Age, Continuous [Mean (Standard Deviation); unit: years] | 70.0 (8.49) | 66.3 (3.06) | 67.8 (5.17)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 1 | 2
  Male | 1 | 2 | 3
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 2 | 3 | 5
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 2 | 3 | 5
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 2 | 3 | 5

OUTCOME MEASURES:

1. Primary Outcome: Determine Changes in Language Performance After Stimulation Sessions
Description: Language performance as assessed at baseline and post-stimulation procedure
Time Frame: Language performance was assessed before and after 2-week intervention and during washout periods
Population: No data were collected for this outcome measure.
Arm/Group | HD-tDCS, Then Sham | Sham, Then HD-tDCS
Number analyzed (Participants) | 0 | 0

2. Secondary Outcome: Determine the Resting State Language Network-level Changes in Left TPC Functional Connectivity.
Description: Language network resting state changes after stimulation procedure
Time Frame: Language network resting state changes were assessed before and after 2-week intervention and during washout periods
Population: No data were collected for this outcome measure.
Arm/Group | HD-tDCS, Then Sham | Sham, Then HD-tDCS
Number analyzed (Participants) | 0 | 0

3. Secondary Outcome: Determine the Neuronal Frequency Distribution and Connectivity Measures Associated With the Left TPC as Assessed by MEG.
Description: Resting-state neuronal frequencies and synchronizations changes after stimulation procedure
Time Frame: Resting-state neuronal frequencies and synchronizations changes were assessed before and after 2-week intervention and during washout periods
Population: No data were collected for this outcome measure.
Arm/Group | HD-tDCS, Then Sham | Sham, Then HD-tDCS
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: Informed consent through study completion, approximately 28 weeks.
Description: Safety Population included all subjects who received at least one intervention.
Groups:
- HD-tDCS: Subjects receive High Dose transcranial Direct Current Stimulation (HD-tDCS) lasting 20 minutes at an electric current intensity of up to 2mA in the left posterior temporo-parietal cortex (TPC). Stimulation sessions are delivered once a day (QD) for a total of 10 sessions over 2 weeks (Monday-Friday).
  Adverse events reported in this group include relevant medical occurrences from the 10 sessions of HD-tDCS through post-intervention follow-up.
  HD-tDCS: High-Dose transcranial Direct Current Stimulation
- Sham: Subjects receive Sham sessions (no electric current) once a day (QD) for a total of 10 sessions over 2 weeks (Monday-Friday).
  Adverse events reported in this group include relevant medical occurrences from the 10 sessions of sham through post-intervention follow-up.
  Sham: Sham sessions (no electric current)
Arm/Group | HD-tDCS | Sham
All-Cause Mortality (participants affected / at risk) | 0/4 | 0/4
Serious Adverse Events (participants affected / at risk) | 1/4 | 0/4
Other Adverse Events (participants affected / at risk) | 2/4 | 1/4
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | HD-tDCS (N=4) | Sham (N=4)
COVID-19 (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | HD-tDCS (N=4) | Sham (N=4)
Bleeding at electrode site (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Erythema at collar bone post MEG (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Headaches (General disorders) | 0 (0) | 1 (1)
Urinary tract infection (Renal and urinary disorders) | 1 (1) | 0 (0)
Fall (Social circumstances) | 1 (1) | 0 (0)
Increased panic attacks (Psychiatric disorders) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2022-05-26): https://cdn.clinicaltrials.gov/large-docs/59/NCT03805659/Prot_000.pdf
  • Statistical Analysis Plan (2023-07-06): https://cdn.clinicaltrials.gov/large-docs/59/NCT03805659/SAP_002.pdf